CLINICAL TRIAL: NCT01097720
Title: Developmental Delay in Children Exposed During Pregnancy to Either Lamotrigine, Sodium Valproate, or Carbamazepine
Brief Title: Developmental Delay in Children Exposed During Pregnancy to Either Lamotrigine,Sodium Valproate, or Carbamazepine
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Lewis B. Holmes, MD, Massachusetts General Hospital
Other Study IDs: 2005P000379
Record Dates: First submitted 2010-03-31; First posted 2010-04-02 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Autism; Developmental Delay; Birth Defects
Keywords: Valproate; Lamotrigine; Carbamazepine; Anticonvulsant; Antiepileptic; Teratogen; Autism; Developmental Delay
MeSH Terms: conditions — Autistic Disorder; Learning Disabilities; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- LTG-exposed: Children exposed to LTG during pregnancy.
- VPA-exposed: Children exposed to VPA during pregnancy.
- CBZ-exposed: Children exposed to CBZ during pregnancy.

SUMMARY:
This study is investigating the neurodevelopmental effects of prenatal exposure to lamotrigine (LTG), sodium valproate (VPA), or carbamazepine (CBZ) monotherapies. The hypotheses to be tested include:

1. Exposure during pregnancy to CBZ, LTG, and VPA, each as monotherapy, is associated with developmental delay with or without signs of autism.
2. Exposure to each drug (CBZ, LTG, and VPA) as monotherapy is associated with an increased rate of occurrence of major malformations.
3. The child with major malformations is more likely to have developmental delay with or without signs of autism than the child who does not have major malformations.
4. The occurrence of adaptive behavior outcomes will show a dose-response relationship with the dose of medication taken by the mother in the first trimester.

The study population includes children 36-83 months of age who were exposed throughout gestation to one of the three drugs of interest, as treatment for maternal seizure disorder.

ELIGIBILITY:
Inclusion Criteria:

* 36-83 months of age
* Prenatal exposure to LTG, VPA, or CBZ monotherapy
* AED was used by mother to suppress seizures
* Mother was enrolled in the North American AED Pregnancy Registry

Exclusion Criteria:

* Exposure during the first trimester to other known teratogens.
* Mother with mental health issues
* Refusal to release medical records to confirm eligibility.

Ages: 36 Months to 83 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children 36-83 months of age, prenatally exposed to LTG, VPA, or CBZ monotherapies, recruited through mothers enrolled in the North American Antiepileptic Drug Pregnancy Registry.
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2005-03; Primary Completion 2010-01 (Actual); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Adaptive Behavior Scores | 36-83 months of age
  Measures of each child's Adaptive Behavior scores as assessed by the Vineland-II Adaptive Behavior Scales, collected when the child was between 36 and 83 months of age.

SECONDARY OUTCOMES:
Presence/Absence of Major Malformations | 36-83 months of age
  Based on interview with mother and review of medical records, determination is made as to whether or not the child had any major malformations at birth.

CONTACTS AND LOCATIONS:
Overall Officials: Lewis B. Holmes, MD, Principal Investigator — Massachusetts General Hospital; Jane Adams, Ph.D., Study Director — University of Massachusetts, Boston
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States